CLINICAL TRIAL: NCT04725240
Title: A Phase 2, Open-Label 20-Week Study to Evaluate the Safety and Efficacy of Setmelanotide in Subjects With Hypothalamic Obesity
Brief Title: Open-Label Study of Setmelanotide in Hypothalamic Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RM-493-030; 2022-004107-32 (EudraCT Number)
Record Dates: First submitted 2021-01-06; First posted 2021-01-26 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Hypothalamic Obesity
MeSH Terms: conditions — Sexual Infantilism | interventions — setmelanotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Setmelanotide (Experimental): Participants received setmelanotide once daily (QD) via SC injection for 16 weeks. All participants initiated treatment with setmelanotide (starting dose being age dependent) and dose escalated up to a maximum dose of 3.0 milligrams (mg) QD.
  Interventions: Drug: Setmelanotide

INTERVENTIONS:
Drug: Setmelanotide — Setmelanotide for SC injection

SUMMARY:
Open-label, single-arm study designed to evaluate the body weight response to setmelanotide administered subcutaneously (SC) daily in participants with hypothalamic obesity (HO).

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be eligible for study participation:

* Participant has documented evidence of HO, including:

  * Recent evidence of hypothalamic injury on magnetic resonance imaging (MRI); AND
  * Diagnosis of craniopharyngioma or other non-malignant brain tumor affecting the hypothalamic region; AND
  * Has undergone surgery, or chemotherapy, or radiation ≥6 months and ≤15 years before Screening.
* Participant has either unilateral hypothalamic lesions or bilateral hypothalamic lesions, as assessed by MRI.
* Obesity, documented by a body mass index (BMI) ≥35 kilograms/square meter (kg/m^2) for participants ≥18 years of age or BMI ≥95th percentile for age and gender for participants 6 to <18 years of age.
* Documented increase in BMI (change from pre-surgery baseline in BMI z-score ≥0.2 for participants <18 years of age or BMI >5% for participants >18 years of age) either during the first 6 months following surgery or within 1 year before surgery AND still present at Screening.
* More than 6 months after the end of post-tumor treatment, including chemotherapy, surgery, or radiation.
* Highly effective contraception throughout the study and for 90 days following the study.
* Ability to communicate well with the Investigator, understand and comply with the requirements of the study, and understand and sign the written informed consent, or, for participants aged <18 years, a parent/legal guardian that can sign.
* If receiving hormone replacement therapy, the dose of such therapy has remained stable for at least 2 months prior to Screening.

Exclusion Criteria:

Participants meeting any of the following criteria are not eligible for study participation:

* Weight gain >5% in the previous 3 months.
* Weight loss ≥2% in the previous 3 months.
* Bariatric surgery or procedure within the last 6 months.
* Diagnosis of severe psychiatric disorders
* Glycated hemoglobin (HbA1c) >10.0% at Screening.
* Current, clinically significant pulmonary, cardiac, or oncologic disease considered severe enough to interfere with the study and/or confound the results.
* Glomerular filtration rate (GFR) <30mL/min/1.73m^2 during Screening.
* Significant dermatologic findings relating to melanoma or pre-melanoma skin lesions.
* History or close family history (parents or siblings) of skin cancer or melanoma
* Participation in any clinical study with an investigational drug/device within 3 months or 5 half-lives, whichever is longer, prior to the first setmelanotide dose.
* Previously enrolled in a clinical study involving setmelanotide or any previous exposure to setmelanotide.
* Inability to comply with QD injection regimen.
* Pregnant and/or breastfeeding, or desiring to become pregnant during this trial.
* Cognitive impairment that, in the Investigator's opinion, precludes participation to the study and completions of study procedures or questionnaires.
* Participant is, in Investigator's opinion, otherwise not suitable to participate in the study.

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Meeker, MD, Study Chair — Rhythm Pharmaceuticals, Inc.
Locations (5):
- United States (5):
  - Rady Children's Hospital, San Diego, California
  - University of Florida, Gainesville, Florida
  - Children's Minnesota, Saint Paul, Minnesota
  - Vanderbilt University School of Medicine, Nashville, Tennessee
  - Seattle Children's Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roth CL, Scimia C, Shoemaker AH, Gottschalk M, Miller J, Yuan G, Malhotra S, Abuzzahab MJ. Setmelanotide for the treatment of acquired hypothalamic obesity: a phase 2, open-label, multicentre trial. Lancet Diabetes Endocrinol. 2024 Jun;12(6):380-389. doi: 10.1016/S2213-8587(24)00087-1. Epub 2024 Apr 30. PMID 38697184

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 19 participants screened, 18 participants were enrolled in the study.
Groups:
- Setmelanotide: Participants received setmelanotide once daily (QD) via subcutaneous (SC) injection for 16 weeks. All participants initiated treatment with setmelanotide (starting dose being age dependent) and dose escalated up to a maximum dose of 3.0 milligrams (mg) QD.
Period: Overall Study
Arm/Group | Setmelanotide
Started | 18
Completed | 16
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set included all participants who received at least 1 dose of setmelanotide and had baseline data.
Groups:
- Setmelanotide: Participants received setmelanotide QD via SC injection for 16 weeks. All participants initiated treatment with setmelanotide (starting dose being age dependent) and dose escalated up to a maximum dose of 3.0 mg QD.
Arm/Group | Setmelanotide
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.0 (5.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/square meter (kg/m^2)] | 37.95 (6.532)
Body Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 102.76 (30.120)
BMI Z-Score [Mean (Standard Deviation); unit: z-score] — The BMI Z-score indicated the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched individuals). A decrease of BMI Z-score indicates a reduction in BMI from Baseline whereas an increase of BMI-Z score indicates an increase in BMI from Baseline. Population: Participants in the Full Analysis Set with available data were analyzed.
  z-score
    number analyzed (Participants) | 13
    (all) | 3.935 (0.9080)
Waist Circumference [Mean (Standard Deviation); unit: centimeters (cm)] | 114.07 (16.354)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With ≥ 5% Reduction in BMI From Baseline After 16 Weeks of Setmelanotide Treatment
Description: BMI was calculated using participant's weight and height assessments, using the following formula: BMI = kg/m^2. Baseline was defined as the most recent measurement prior to the first administration of study drug.
Time Frame: Baseline to 16 weeks
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Setmelanotide
Number analyzed (Participants) | 18
percentage of participants | 88.9 [69.0 to 98.0]
Statistical Analysis 1: Comparison: Setmelanotide; Test type: Other; p < 0.0001, One-sided exact binomial test — Threshold for significance at 0.001 level

2. Secondary Outcome: Composite Percentage of Participants Aged ≥6 to <18 Years With ≥0.2 Reduction of BMI Z-Score or Participants Aged ≥18 Years With 5% Reduction of Body Weight From Baseline After 16 Weeks of Setmelanotide Treatment
Description: For participants aged ≥6 to <18 years, a participant's BMI Z-score was considered for the analysis; for participants ≥18 years, a participant's body weight (kg) was considered for the analysis. BMI was calculated using participant's weight and height assessments, using the following formula: BMI = kg/m^2. The BMI Z-score indicated the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched individuals). A decrease of BMI Z-score indicates a reduction in BMI from Baseline whereas an increase of BMI-Z score indicates an increase in BMI from Baseline. Baseline was defined as the most recent measurement prior to the first administration of study drug.
Time Frame: Baseline to Week 16
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Setmelanotide
Number analyzed (Participants) | 18
percentage of participants | 88.9 [69.0 to 98.0]
Statistical Analysis 1: Comparison: Setmelanotide; Test type: Other; p < 0.0001, One-sided exact binomial test — Threshold for significance at 0.001 level

3. Secondary Outcome: Percentage of Participants Aged ≥6 to <18 Years With ≥0.2 Reduction of BMI Z-Score From Baseline After 16 Weeks of Setmelanotide Treatment
Description: BMI was calculated using participant's weight and height assessments, using the following formula: BMI = kg/m^2. The BMI Z-score indicated the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched individuals). A decrease of BMI Z-score indicates a reduction in BMI from Baseline whereas an increase of BMI-Z score indicates an increase in BMI from Baseline. Baseline was defined as the most recent measurement prior to the first administration of study drug.
Time Frame: Baseline to 16 weeks
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Setmelanotide
Number analyzed (Participants) | 13
percentage of participants | 92.3 [68.4 to 99.6]
Statistical Analysis 1: Comparison: Setmelanotide; Test type: Other; p < 0.0001, One-sided exact binomial test — Threshold for significance at 0.001 level

4. Secondary Outcome: Percentage of Participants Aged ≥18 Years With ≥5% Reduction of Body Weight From Baseline After 16 Weeks of Setmelanotide Treatment
Description: Baseline was defined as the most recent measurement prior to the first administration of study drug.
Time Frame: Baseline to Week 16
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Setmelanotide
Number analyzed (Participants) | 5
percentage of participants | 80.0 [34.3 to 99.0]
Statistical Analysis 1: Comparison: Setmelanotide; Test type: Other; p < 0.0001, One-sided exact binomial test — Threshold for significance at 0.001 level

5. Secondary Outcome: Change From Baseline in Waist Circumference in Participants Aged ≥18 Years After 16 Weeks of Setmelanotide Treatment
Description: Waist circumference was measured after participants had fasted for at least 8 hours and at approximately the same time at each visit. Baseline was defined as the most recent measurement prior to the first administration of study drug.
Time Frame: Baseline, Week 16
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Setmelanotide
Number analyzed (Participants) | 4
cm | -10.275 (4.2272)

6. Secondary Outcome: Change From Baseline in Daily Hunger Questionnaire Score in Participants Aged <12 Years After 16 Weeks of Setmelanotide Treatment
Description: Daily Hunger Questionnaire for participants <12 years of age: Three aspects of hunger (average hunger in the last 24 hours, most/worst hunger in the last 24 hours, and morning hunger) were assessed daily using a pictorial (smiley face) version of the Likert rating scale with scores from 0 to 4, with 0 = not hungry at all and 4 = hungriest possible. Responses were recorded in the electronic diary. Each of the 3 items (average hunger, most/worst hunger, and morning hunger) was scored separately and averaged to calculate a total score ranging from 0 (not hungry at all) to 4 (hungriest possible) with higher score indicating more hunger. Baseline daily hunger score was calculated as the average of 7 days prior to Baseline visit.
Time Frame: Baseline, Week 16
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Setmelanotide
Number analyzed (Participants) | 5
units on a scale | -1.490 (1.2126)

7. Secondary Outcome: Change From Baseline in Daily Hunger Questionnaire Scores in Participants Aged ≥12 Years After 16 Weeks of Setmelanotide Treatment
Description: Daily Hunger Questionnaire for participants ≥12 years of age: Three aspects of hunger (average hunger in the last 24 hours, most/worst hunger in the last 24 hours, and morning hunger) were assessed daily using a numeric rating score for each from 0 to 10, with 0 = not hungry at all and 10 = hungriest possible. The responses to the Daily Hunger Questionnaire were recorded in the electronic diary. Baseline daily hunger score was calculated as the average of 7 days prior to Baseline visit.
Time Frame: Baseline, Week 16
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Setmelanotide
Number analyzed (Participants) | 11
units on a scale
  Most hunger | -2.922 (2.2851)
  Average hunger | -3.122 (1.9999)
  Morning hunger | -2.717 (1.9393)

8. Secondary Outcome: Number of Participants With Shift From Baseline in Global Hunger Questionnaire Score to Week 16 in Participants Aged < 12 Years
Description: Parents or caregivers of participants <12 years old answered the Caregiver Reported Global Hunger Question for participants who were <12 years old. The following question was asked: How hungry is your child acting now? Possible responses were: Not hungry at all; A little hungry; Moderately hungry; and Extremely hungry. Baseline was defined as the most recent measurement prior to the first administration of study drug.
Time Frame: Baseline, Week 16
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Setmelanotide
Number analyzed (Participants) | 5
Participants
  Not hungry at all (Baseline) - Not hungry at all (Week 16) | 0
  A little hungry (Baseline) - Not hungry at all (week 16) | 0
  Moderately hungry (Baseline) - Not hungry at all (Week 16) | 0
  Extremely hungry (Baseline) - Not hungry at all (Week 16) | 2
  Not hungry at all (Baseline) - A little hungry (Week 16) | 0
  A little hungry (Baseline) - A little hungry (Week 16) | 0
  Moderately hungry (Baseline) - A little hungry (Week 16) | 1
  Extremely hungry (Baseline) - A little hungry (Week 16) | 2
  Not hungry at all (Baseline) - Moderately hungry (Week 16) | 0
  A little hungry (Baseline) - Moderately hungry (Week 16) | 0
  Moderately hungry (Baseline) - Moderately hungry (Week 16) | 0
  Extremely hungry (Baseline) - Moderately hungry (Week 16) | 0
  Not hungry at all (Baseline) - Extremely hungry (Week 16) | 0
  A little hungry (Baseline) - Extremely hungry (Week 16) | 0
  Moderately hungry (Baseline) - Extremely hungry (Week 16) | 0
  Extremely hungry (Baseline) - Extremely hungry (Week 16) | 0

9. Secondary Outcome: Number of Participants With Shift From Baseline in Global Hunger Questionnaire Score to Week 16 in Participants Aged ≥12 Years
Description: Global Hunger Questionnaire for participants ≥12 years of age. The following question was asked: Overall, how would you rate the hunger you experience now? Possible responses were: No hunger; Mild hunger; Moderate hunger; and Severe hunger. Baseline was defined as the most recent measurement prior to the first administration of study drug.
Time Frame: Baseline, Week 16
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Setmelanotide
Number analyzed (Participants) | 11
Participants
  No hunger (Baseline) - No hunger (Week 16) | 0
  Mild hunger (Baseline) - No hunger (Week 16) | 1
  Moderate hunger (Baseline) - No hunger (Week 16) | 3
  Severe hunger (Baseline) - No hunger (Week 16) | 0
  No hunger (Baseline) - Mild hunger (Week 16) | 1
  Mild hunger (Baseline) - Mild hunger (Week 16) | 0
  Moderate hunger (Baseline) - Mild hunger (Week 16) | 3
  Severe hunger (Baseline) - Mild hunger (Week 16) | 2
  No hunger (Baseline) - Moderate hunger (Week 16) | 0
  Mild hunger (Baseline) - Moderate hunger (Week 16) | 0
  Moderate hunger (Baseline) - Moderate hunger (Week 16) | 1
  Severe hunger (Baseline) - Moderate hunger (Week 16) | 0
  No hunger (Baseline) - Severe hunger (Week 16) | 0
  Mild hunger (Baseline) - Severe hunger (Week 16) | 0
  Moderate hunger (Baseline) - Severe hunger (Week 16) | 0
  Severe hunger (Baseline) - Severe hunger (Week 16) | 0

10. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence or clinically significant worsening of an existing condition associated with the use of a drug in humans, whether or not considered drug related. An AE (also referred to as an adverse experience) could be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, without any judgment about causality.
Time Frame: From first dose of study drug up to Day 141
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Setmelanotide
Number analyzed (Participants) | 18
Participants | 18

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Day 141
Description: Participants in the Safety Analysis Set were analyzed.
Arm/Group | Setmelanotide
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 1/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Setmelanotide (N=18)
Clostridium difficile colitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Setmelanotide (N=18)
Fatigue (General disorders) | 3
Injection site pain (General disorders) | 3
Injection site pruritus (General disorders) | 2
Pain (General disorders) | 2
Pyrexia (General disorders) | 2
Injection site erythema (General disorders) | 1
Injection site induration (General disorders) | 1
Injection site swelling (General disorders) | 1
Erection increased (Reproductive system and breast disorders) | 3/11 — This denominator includes only the male participants in the group (N = 11).
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Conversion disorder (Psychiatric disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood uric acid increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Weight decreased (Investigations) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Radius fracture (Injury, poisoning and procedural complications) | 1
Type V hyperlipidaemia (Congenital, familial and genetic disorders) | 1
Headache (Nervous system disorders) | 2
Balance disorder (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Speech disorder (Nervous system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Nausea (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Portal hypertensive gastropathy (Gastrointestinal disorders) | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 6
Acne (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 1
COVID-19 (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 2
Administration site cellulitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Staphylococcal abscess (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information regarding setmelanotide supplied by Rhythm to the investigator is privileged and confidential information. The investigator agrees to use this information to accomplish the study and will not use it for other purposes without consent from Rhythm. The information obtained from the clinical study will be used towards the development of setmelanotide and may be disclosed to regulatory authority(ies), other investigators, corporate partners, or consultants as required.

DOCUMENTS (2):
  • Study Protocol (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT04725240/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT04725240/SAP_001.pdf